CLINICAL TRIAL: NCT01127659
Title: Effect of Hypogonadotrophic Hypogonadism and Treatment With Testosterone on Insulin Sensitivity, Inflammation, Body Composition and Sexual Function in Obese and Type 2 Diabetic Men
Brief Title: Testosterone Replacement in Men With Diabetes and Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIH testosterone grant; R01DK075877 (NIH)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-10

CONDITIONS: Hypogonadism
Keywords: diabetes; hypogonadism; obesity; testosterone; insulin sensitivity; inflammation
MeSH Terms: conditions — Hypogonadism; Diabetes Mellitus; Obesity; Insulin Resistance; Inflammation | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- diabetes with HH-active (Active Comparator): Subjects with diabetes and hypogonadotropic hypogonadism. They will be randomized to testosterone intervention.
  Interventions: Drug: testosterone
- diabetes with normal testosterone (No Intervention): Eugonadal subjects with diabetes. They will not be treated
- obese with HH-active (Active Comparator): Obese non-diabetic men hypogonadotropic hypogonadism. They will be randomized to testosterone intervention.
  Interventions: Drug: testosterone
- obese with normal testosterone (No Intervention): Eugonadal non-diabetic obese subjects. They will not be treated
- Diabetes with HH-placebo (Placebo Comparator): Subjects with diabetes and hypogonadotropic hypogonadism. They will be randomized to placebo.
  Interventions: Drug: placebo
- Obese with HH-placebo (Placebo Comparator): Obese non-diabetic men hypogonadotropic hypogonadism. They will be randomized to placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: testosterone — intramuscular every 2 weeks
  Arms: diabetes with HH-active; obese with HH-active
Drug: placebo — saline intramuscular every 2 weeks
  Arms: Diabetes with HH-placebo; Obese with HH-placebo

SUMMARY:
The purpose of this study is to examine the effect of having testosterone deficiency in men with diabetes and with obesity. The study will also evaluate the effect of testosterone therapy. This will be done by comparing the changes in several body response indicators following treatment with testosterone in diabetic or obese-non diabetic men with low testosterone levels and comparing them to diabetic or obese-non diabetic men with low testosterone who are not treated with testosterone.

DETAILED DESCRIPTION:
Hypogonadotropic hypogonadism (HH) occurs in approximately one-third of obese and type 2 diabetic men. Considering that there are 24 million diabetic and 100 million obese people, of which half are males, obesity and type 2 diabetes potentially constitute the major cause of hypogonadism in the population. We hypothesize that 1) HH in obese and type 2 diabetic men is associated with decreased insulin sensitivity, increased fat tissue mass, decreased lean body mass, increased inflammatory and oxidative stress, impaired sexual function and depressed mood as compared to diabetic and obese men with normal testosterone concentrations; and that 2) testosterone replacement for 24 weeks in men with HH leads to an improvement in these parameters. Our proposed study would be the first prospective, randomized trial to comprehensively evaluate the effect of HH on insulin sensitivity, body composition, inflammatory and oxidative indices in obese and type 2 diabetic subjects and the effect of six months of T replacement on these parameters. The study will have 2 arms (obese and type 2 diabetic arm) with 120 subjects in Diabetes arm and 80 subjects in obese arm. Half of men in each arm will have HH and half men will have normal testosterone concentrations(eugonadal men). Insulin sensitivity will be assessed by hyperinsulinemic-euglycemic clamps. Subcutaneous fat mass and lean body mass will be measured by DEXA and intra-abdominal (visceral) fat mass by MRI. All subjects will undergo hyperinsulinemic-euglycemic clamp, MRI, DEXA and give blood and urine samples (for measurement of inflammatory and oxidative stress) at baseline. Men with HH will then be randomized to receive testosterone or placebo gel for a total of 24 weeks. These men will undergo hyperinsulinemic-euglycemic clamps and give blood and urine samples for inflammation and oxidative stress at 4 weeks and 24 weeks. MRI and DEXA examinations will be carried out at 24 weeks again in men with HH. The primary endpoint of the study is to define a difference in whole body glucose uptake during hyperinsulinemic-euglycemic clamps between hypogonadal and eugonadal diabetes patients at baseline and an increase in glucose uptake in HH subjects after treatment with testosterone for 24 weeks. 30 subjects per group(testosterone and placebo gel each) will provide adequate power (0.8) to detect a significant difference of 10% in whole body glucose uptake. Therefore there will be 60 men with HH in each arm in diabetes group. For baseline comparisons, 60 men with normal testosterone concentrations will also be needed in each arm. We will recruit 40 obese patients in each arm. Thus there will be 120 diabetic men and 80 obese men in the study.

ELIGIBILITY:
Inclusion Criteria:

* T2D arm: Males with age 30-65 years
* Obese non-diabetic arm: Obese non-diabetic males with age 30-65 years

Exclusion Criteria:

1)Coronary event or procedure(myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous twelve weeks; 2) PSA > 4ng/ml; 3)Hemoglobin A1c > 8%; 4)h/o prostate carcinoma; 5)Hepatic disease (transaminase > 3 times normal) or cirrhosis; 6)Renal impairment (defined as GFR<30); 7)HIV or Hepatitis C positive status; 9)Participation in any other concurrent clinical trial; 10)Any other life-threatening, non-cardiac disease; 11)Use of over the counter health supplements which contain androgens; 12)Use of an investigational agent or therapeutic regimen within 30 days of study; 13)prostate nodule or severe enlargement on digital rectal examination; 14)Use of testosterone currently or in the past 4 months; 15)Hematocrit > 50%; 16)History of untreated severe obstructive sleep apnea(defined as apnea-hypopnea index ≥30); 17)symptoms suggestive of severe BPH; 18)Congestive heart failure, class III or IV; 20)Known to have anemia secondary to iron, B12 or folic acid deficiency; 21)bone marrow disorder such as myelodysplasia or aplastic anemia; 22) currently suffering from symptomatic depression, with or without treatment; 23) history of severe depression in the past which needed hospitalization; 24)currently suffering from foot ulcer, significant periodontal disease or any other chronic infectious condition; 25)planning to have children. 26) Subjects on testosterone or with testosterone replacement in the past 4 months will be excluded.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-05; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MBBS, Principal Investigator — SUNY at Buffalo
Locations (1):
- 115 Flint Road, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghanim H, Dhindsa S, Batra M, Green K, Abuaysheh S, Kuhadiya ND, Makdissi A, Chaudhuri A, Sandhu S, Dandona P. Testosterone Increases the Expression and Phosphorylation of AMP Kinase alpha in Men With Hypogonadism and Type 2 Diabetes. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1169-75. doi: 10.1210/clinem/dgz288. PMID 31858126
- [Derived] Ghanim H, Dhindsa S, Batra M, Green K, Abuaysheh S, Kuhadiya ND, Makdissi A, Chaudhuri A, Dandona P. Effect of Testosterone on FGF2, MRF4, and Myostatin in Hypogonadotropic Hypogonadism: Relevance to Muscle Growth. J Clin Endocrinol Metab. 2019 Jun 1;104(6):2094-2102. doi: 10.1210/jc.2018-01832. PMID 30629183
- [Derived] Dhindsa S, Ghanim H, Batra M, Kuhadiya ND, Abuaysheh S, Sandhu S, Green K, Makdissi A, Hejna J, Chaudhuri A, Punyanitya M, Dandona P. Insulin Resistance and Inflammation in Hypogonadotropic Hypogonadism and Their Reduction After Testosterone Replacement in Men With Type 2 Diabetes. Diabetes Care. 2016 Jan;39(1):82-91. doi: 10.2337/dc15-1518. Epub 2015 Nov 29. PMID 26622051

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes With HH: Testosterone: active drug diabetes arm
  testosterone: intramuscular every 2 weeks
- Diabetes With HH: Placebo: placebo diabetes arm
  placebo: saline intramuscular every 2 weeks
- Obese Testosterone: active drug obese arm
  testosterone: intramuscular every 2 weeks
- Obese Placebo: placebo obese arm
  placebo: saline intramuscular every 2 weeks
- Eugonadal Diabetes; Eugonadal Obese: no intervention. Only baseline data collected
Period: Overall Study
Arm/Group | Diabetes With HH: Testosterone | Diabetes With HH: Placebo | Obese Testosterone | Obese Placebo | Eugonadal Diabetes | Eugonadal Obese
Started | 22 | 22 | 12 | 10 | 50 | 21
Completed | 20 | 14 | 10 | 6 | 50 | 21
Not Completed | 2 | 8 | 2 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diabetes With HH: Testosterone: active drug diabetes hypogonadal arm
  testosterone: intramuscular every 2 weeks
- Obese With HH: Testosterone: active drug obese hypogonadal arm
  testosterone: intramuscular every 2 weeks
- Obese With HH: Placebo: placebo obese hypogonadal arm
  placebo: saline intramuscular every 2 weeks
- Diabetes With HH: Placebo: placebo diabetes hypogonadal arm
  placebo: saline intramuscular every 2 weeks
- Eugonadal Diabetes: diabetic men with normal testosterone
- Eugonadal Obese: obese non-diabetic men with normal testosterone
- Total: Total of all reporting groups
Arm/Group | Diabetes With HH: Testosterone | Obese With HH: Testosterone | Obese With HH: Placebo | Diabetes With HH: Placebo | Eugonadal Diabetes | Eugonadal Obese | Total
Number analyzed (Participants) | 22 | 12 | 10 | 22 | 50 | 21 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 12 | 10 | 22 | 50 | 21 | 137
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7) | 46 (9) | 53 (7) | 54 (9) | 52 (9) | 50 (8) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 22 | 12 | 10 | 22 | 50 | 21 | 137
Region of Enrollment [Number; unit: participants]
  United States | 22 | 12 | 10 | 22 | 50 | 21 | 137

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: measured by HE clamps (baseline and 6 mths)
Time Frame: baseline to 6 months
Population: Glucose infusion rate in HE clamps was measured
Measure: Mean (Standard Deviation); unit: mg/kg fat free mass/min
Groups:
- Diabetes With HH: Testosterone: active drug diabetes hypogonadal arm
  testosterone: intramuscular every 2 weeks
  Glucose infusion rate: 6.5+/-4.0 mg/kg fat-free mass/min
- Eugonadal Diabetes: diabetic men with normal testosterone. these participants did not contribute to the assessment at 6 months because they did not undergo the intervention
- Eugonadal Obese: obese non-diabetic men with normal testosterone. these participants did not contribute to the assessment at 6 months because they did not undergo the intervention
Arm/Group | Diabetes With HH: Testosterone | Diabetes With HH: Placebo | Obese With HH: Testosterone | Obese With HH: Placebo | Eugonadal Diabetes | Eugonadal Obese
Number analyzed (Participants) | 20 | 14 | 10 | 6 | 50 | 21
mg/kg fat free mass/min
  baseline | 6.66 (4.36) | 5.12 (2.79) | 11.37 (8.83) | 12.93 (5.16) | 10.29 (5.55) | 12.30 (5.96)
  6 months: number analyzed (Participants) | 20 | 14 | 10 | 6 | 0 | 0
  6 months | 8.73 (4.27) | 5.06 (3.62) | 12.96 (7.11) | 14.57 (1.71) |  |

2. Secondary Outcome: Body Composition
Description: Body composition using Total body fat mass (kg)
Time Frame: baseline to 6 months
Population: Body composition using Total body fat mass (kg)
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Eugonadal Diabetes; Eugonadal Obese: no intervention. these participants did not contribute to the assessment at 6 months because they did not undergo the intervention.
Arm/Group | Diabetes With HH: Testosterone | Diabetes With HH: Placebo | Obese Testosterone | Obese Placebo | Eugonadal Diabetes | Eugonadal Obese
Number analyzed (Participants) | 20 | 14 | 10 | 6 | 50 | 21
kg
  Baseline | 44.5 (13.7) | 44.5 (15.0) | 50.2 (9.5) | 48.8 (10.4) | 34.0 (12.0) | 40.2 (12.4)
  24 WEEKS: number analyzed (Participants) | 20 | 14 | 10 | 6 | 0 | 0
  24 WEEKS | 42.1 (12.5) | 45.4 (14.4) | 46.4 (11.7) | 48.4 (11.2) |  |

ADVERSE EVENTS:
Arm/Group | Diabetes With HH: Testosterone | Diabetes With HH: Placebo | Obese With HH: Testosterone | Obese With HH: Placebo | Eugonadal Diabetes | Eugonadal Obese
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/12 | 0/10 | 0/50 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/12 | 0/10 | 0/50 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes